CLINICAL TRIAL: NCT02478879
Title: An Open-label Crossover Study to Determine the Patient Preference Between ZP-PTH Patches and Forteo Pens After Daily Treatment for 14 Days in Women 55-85 Years of Age
Brief Title: A Study to Determine the Patient Preference Between Zosano Pharma Parathyroid Hormone (ZP-PTH) Patch and Forteo Pen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zosano Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-2015-005
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Parathyroid Hormone; Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZP-PTH Patch (Experimental): Intradermal microneedle patch coated with 40 mcg of PTH, applied intracutaneously to the abdomen daily for 30 minutes, 14 days of treatment
  Interventions: Drug: ZP-PTH
- FORTEO(R) Pen (Active Comparator): Marketed FORTEO 20 mcg, administered daily as a subcutaneous injection to the abdomen or thigh for 14 days of treatment.
  Interventions: Drug: FORTEO

INTERVENTIONS:
Drug: ZP-PTH — Patch applied daily for 30 minutes, 14 days
  Other Names: PTH; parathyroid hormone; teriparatide
  Arms: ZP-PTH Patch
Drug: FORTEO — Subcutaneous injection administration daily for 14 days
  Other Names: PTH; FORSTEO; teriparatide
  Arms: FORTEO(R) Pen

SUMMARY:
The purpose of this study is to determine which of two delivery methods of Parathyroid Hormone (PTH) is preferred by patients after 14 days of use for each.

DETAILED DESCRIPTION:
The purpose of this study is to determine which of two delivery methods of PTH is preferred by patients after 14 days of use for each. Patient preference will be determined by means of patient questionnaires at the end of each treatment period and a final questionnaire after both treatment periods are complete. Adverse events will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal with prior diagnosis of osteoporosis

Exclusion Criteria:

* Significant health issue
* previous use of teriparatide
* History of Paget's disease

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall Preference | 28 days
  The fraction of subjects expressing an overall preference for each treatment based on a 4 point scale

SECONDARY OUTCOMES:
Safety (adverse events) | 28 days
  incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Coleman, DO, Principal Investigator — Convance
Locations (1):
- Covance Daytona Beach Clinical Research Unit, Daytona Beach, Florida, United States